CLINICAL TRIAL: NCT01891396
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of a Single Injection Cross-Linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide (Cingal) to Provide Symptomatic Relief of Osteoarthritis of the Knee
Brief Title: Cingal Study for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cingal 13-01
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Hyaluronic acid; HA Injection; Steroid Injection; Knee injection
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and Outcomes Assessor were blinded to treatment
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (Placebo Comparator): Single injection of 0.9% saline supplied as a 4 milliliter (mL) unit dose in a 5mL glass syringe
  Interventions: Device: Saline
- Hyaluronic Acid and TH (Cingal®) (Experimental): Single injection of sodium hyaluronate with triamcinolone hexacetonide (TH) supplied as a 4 milliliter (mL) unit dose in a 5 mL glass syringe
  Interventions: Device: Hyaluronic Acid and TH (Cingal®)
- Hyaluronic Acid (Monovisc®) (Active Comparator): Single injection of sodium hyaluronate supplied as a 4 milliliter (mL) unit dose in a 5 mL glass syringe
  Interventions: Device: Hyaluronic Acid (Monovisc®)

INTERVENTIONS:
Device: Hyaluronic Acid and TH (Cingal®) — Injection into knee
  Other Names: Cingal®
  Arms: Hyaluronic Acid and TH (Cingal®)
Device: Hyaluronic Acid (Monovisc®) — Injection into knee
  Other Names: Monovisc®
  Arms: Hyaluronic Acid (Monovisc®)
Device: Saline — Saline placebo packaged to look identical to comparator syringes. Injection into knee.
  Arms: Saline

SUMMARY:
The purpose of this study is to see if a single injection of Cingal into the knee provides safe relief of pain caused by osteoarthritis.

DETAILED DESCRIPTION:
This study compared three groups of subjects. Group One received a single injection of Cingal (Hyaluronic Acid plus Triamcinolone Hexacetonide). Group Two received a single injection of Monovisc (Hyaluronic Acid). Group Three received a single injection of saline as a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 40 - 75 years old with a Body Mass Index (BMI)≤ 40 kg/m2
* Subject has Kellgren-Lawrence (K-L) severity grade I, II, or III in the index knee as determined by X-Ray. Contralateral knee: K-L severity grade 0, I, or II.

Exclusion Criteria:

* Subject received an intra-articular (IA) injection of Hyaluronic Acid (HA) and/or steroid in either knee within 6 months of signing the informed consent form (ICF).
* Subject had an arthroscopy of either knee within 3 months of signing the informed consent form (ICF).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Hangody, MD, Principal Investigator — Uzsoki Hospital
Locations (27):
- Bulgaria (5):
  - Orthopaedics Clinic Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Clinic of Orthopaedics and Traumatology, University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna", Sofia
  - Consultative Outpatients' Medical Office for Rheumatologic Diseases, Sofia
  - Department of Orthopaedics and Traumatology Multiprofile Hospital for Active Treatment Lyulin Hospital, Sofia
  - Department of Orthopaedics Traumatology - Tokuda Hospital Sofia, Sofia
- Canada (4):
  - Red Deer Regional Hospital Center, Red Deer, Alberta
  - Deakon Medicine Professional Corporation, Oakville, Ontario
  - Sports Medicine Specialists, Toronto, Ontario
  - QEII Health Sciences, Halifax
- Czechia (5):
  - Revmacentrum MUDr. Moster, s.r.o., Brno
  - Faculty Hospital Plzen, Pilsen
  - Institute of Rheumatology, Prague
  - Thomayer Hospital Rheumatology Department, Prague
  - Medical Plus s.r.o., Uherské Hradiště
- Hungary (7):
  - Health Center of Downtown-Lipotvaros, Orthopedic Outpatient Clinic, Budapest
  - Semmelweis Egyetem Orthopaedic Clinic, Budapest
  - Uzsoki Hospital, Department of Traumatology, Budapest
  - Petz Aladar County Teachin Hospital, Traumatology, Orthopaedics and Hand Surgery Centre, Győr
  - Jutrix Medical LLC, Kecskemét
  - Medidea Bt., Kiskunfélegyháza
  - G&V Pharma-Med Bt., Makó
- Poland (6):
  - Osteo-Medic s.c., Bialystok
  - NZOZ Medi SPATX, Gliwice
  - ARTIMED Niepubliczny Zakład Opieki Zdrowotnej, Kielce
  - CenterMed Krakow Sp. x. o.o., Krakow
  - Radlinski Regional Centre of Orthopeadics and Rehabilitation of Locomotor Organs, Lodz
  - Wojewódzki Zespół Reumatologiczny im. Dr Jadwigi Titz-Kosko, Sopot

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hangody L, Szody R, Lukasik P, Zgadzaj W, Lenart E, Dokoupilova E, Bichovsk D, Berta A, Vasarhelyi G, Ficzere A, Hangody G, Stevens G, Szendroi M. Intraarticular Injection of a Cross-Linked Sodium Hyaluronate Combined with Triamcinolone Hexacetonide (Cingal) to Provide Symptomatic Relief of Osteoarthritis of the Knee: A Randomized, Double-Blind, Placebo-Controlled Multicenter Clinical Trial. Cartilage. 2018 Jul;9(3):276-283. doi: 10.1177/1947603517703732. Epub 2017 May 23. PMID 28535076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 594 potential subjects were screened for the study. 226 subjects were screen failures. 368 subjects were randomized into Cingal 13-01 and all received the study injection.
Pre-assignment Details: The most common reason that subjects were excluded before being assigned to a study group (screen failures) was that enrollment target had been reached while subjects were in screening process. Other reasons for screen failure included radiological failures; Kellgren-Lawrence grade not meeting eligibility in the index or contralateral knee.
Groups:
- Hyaluronic Acid and TH (Cingal®): Single injection of sodium hyaluronate with triamcinolone hexacetonide (TH) supplied as a 4 milliliter (mL) unit dose in a 5 mL glass syringe
  Hyaluronic Acid and TH
- Hyaluronic Acid (Monovisc®): Single injection of sodium hyaluronate supplied as a 4 milliliter (mL) unit dose in a 5 mL glass syringe
  Hyaluronic Acid
- Saline: Single injection of 0.9% saline supplied as a 4 milliliter (mL) unit dose in a 5mL glass syringe
  Saline: Saline placebo packaged to look identical to comparator syringes.
Period: Overall Study
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®) | Saline
Started | 149 | 150 | 69
Received Study Injection | 149 | 150 | 69
Completed | 145 | 145 | 66
Not Completed | 4 | 5 | 3
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hyaluronic Acid and TH (Cingal®): Single injection of sodium hyaluronate with triamcinolone hexacetonide (TH) supplied as a 4 mL unit dose in a 5 mL glass syringe
  Hyaluronic Acid and TH
- Hyaluronic Acid (Monovisc®): Single injection of sodium hyaluronate supplied as a 4 mL unit dose in a 5 mL glass syringe
  Hyaluronic Acid
- Saline: Single injection of 0.9% saline supplied as a 4 mL unit dose in a 5mL glass syringe
  Saline: Saline placebo packaged to look identical to comparator syringes.
- Total: Total of all reporting groups
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®) | Saline | Total
Number analyzed (Participants) | 149 | 150 | 69 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.52 (8.39) | 59.19 (8.62) | 58.03 (9.02) | 58.30 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 99 | 51 | 247
  Male | 52 | 51 | 18 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 149 | 149 | 69 | 367
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Saline (ITT)
Description: The change in knee pain from baseline to 12 weeks as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Saline group (ITT population). The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 12 Weeks
Population: Intent To Treat (ITT) Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®) | Saline
Number analyzed (Participants) | 149 | 150 | 69
score on a scale | -40.2 (1.7) | -36.1 (1.6) | -31.0 (2.3)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0099, ANOVA

2. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Monovisc® (ITT)
Description: The change in knee pain from baseline to 1 week post treatment as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Monovisc® group (ITT population). The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 1 Week
Population: Intent To Treat (ITT) Population comparing Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 149 | 150
score on a scale | -34.6 (20.8) | -29.6 (21.4)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0367, ANOVA

3. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Monovisc® (ITT)
Description: The change in knee pain from baseline to 3 weeks as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Monovisc® group (ITT population). The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the change from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 3 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 149 | 150
score on a scale | -40.1 (20.1) | -34.9 (21.7)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0289, ANOVA

4. Secondary Outcome: OMERACT-OARSI Responder Index Comparing Cingal® to Saline (ITT)
Description: The post treatment Responder Rate at 12 weeks is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder. The criteria for response are (1) improvement in pain or physical function ≥50% and an absolute change ≥20 mm; or (2) improvement of ≥20% with an absolute change ≥10 mm in at least two of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome.
Time Frame: 12 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Number; unit: percentage of subjects
Groups:
- Hyaluronic Acid and TH (Cingal®): Single injection of sodium hyaluronate with triamcinolone hexacetonide (TH) supplied as a 4 mL unit dose in a 5 mL glass syringe
  Hyaluronic Acid and TH (Cingal®): Injection into knee
- Saline: Single injection of 0.9% saline supplied as a 4 mL unit dose in a 5mL glass syringe
  Saline: Saline placebo packaged to look identical to comparator syringes. Injection into knee.
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 149 | 69
percentage of subjects | 92.0 | 81.9
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0141, ANOVA

5. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Saline (ITT)
Description: The change from baseline to 12 weeks in the Patient Global Assessment (PGA) comparing the Cingal® and Saline arms (ITT population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 mm = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 12 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 149 | 69
score on a scale | -36.5 (1.6) | -25.3 (2.4)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0002, ANOVA

6. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Monovisc® (ITT)
Description: The change from baseline to 1 week in the Patient Global Assessment (PGA) comparing the Cingal® and Monovisc® arms (ITT population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 1 Week
Population: Intent To Treat (ITT) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Hyaluronic Acid and TH (Cingal®): Single injection of sodium hyaluronate with triamcinolone hexacetonide (TH) supplied as a 4 mL unit dose in a 5 mL glass syringe
- Hyaluronic Acid (Monovisc®): Single injection of sodium hyaluronate supplied as a 4 mL unit dose in a 5 mL glass syringe
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 149 | 150
score on a scale | -32.8 (23.3) | -24.7 (22.6)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0533, ANOVA

7. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Monovisc® (ITT)
Description: Mean change from baseline to 3 weeks in the Patient Global Assessment (PGA) comparing the Cingal® and Monovisc® arms (ITT population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 3 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 149 | 150
score on a scale | -37.7 (23.9) | -32.1 (23.7)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0323, ANOVA

8. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Saline (ITT)
Description: Mean change in knee pain from baseline to 26 weeks as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Saline group. The WOMAC Pain Score is a validated 100mm visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 149 | 69
score on a scale | -41.1 (1.7) | -31.4 (2.4)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0072, ANOVA

9. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Saline (ITT)
Description: Mean change from baseline to 12 weeks in the Evaluator Global Assessment comparing the Cingal® and Saline arms (ITT population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 12 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 149 | 69
score on a scale | -36.8 (1.5) | -27.2 (2.8)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0030, ANOVA

10. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Monovisc® (ITT)
Description: Mean change from baseline to 1 week in the Evaluator Global Assessment comparing the Cingal® and Monovisc® arms (ITT population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 1 Week
Population: Intent To Treat (ITT) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 149 | 150
score on a scale | -31.7 (20.4) | -26.9 (19.7)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0440, ANOVA

11. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Monovisc® (ITT)
Description: Mean change from baseline to 3 weeks in the Evaluator Global Assessment comparing the Cingal® and Monovisc® arms (ITT population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 3 Week
Population: Intent To Treat (ITT) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 149 | 150
score on a scale | -37.5 (21.0) | -32.6 (21.3)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0579, ANOVA

12. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Saline (ITT)
Description: Mean change from baseline to 26 weeks in the Patient Global Assessment (PGA) comparing the Cingal® and Saline arms (ITT population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 149 | 69
score on a scale | -37.0 (1.5) | -26.3 (2.5)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0005, ANOVA

13. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Saline (ITT)
Description: Mean change from baseline to 26 weeks in the Evaluator Global Assessment comparing the Cingal® and Saline arms (ITT population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 26 Weeks
Population: Intent To Treat (ITT) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 149 | 69
score on a scale | -37.8 (1.5) | -28.7 (2.8)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0046, ANOVA

14. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Saline (PP)
Description: The change in knee pain from baseline to 12 weeks as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Saline group (PP population). The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 12 Weeks
Population: Per Protocol (PP) Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®) | Saline
Number analyzed (Participants) | 137 | 135 | 63
score on a scale | -40.3 (1.4) | -35.9 (1.62) | -32.2 (2.2)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0029, ANOVA

15. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Monovisc® (PP)
Description: Mean change in knee pain from baseline to 1 week as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Monovisc® group (PP population). The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 1 Week
Population: Per Protocol (PP) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 136 | 135
score on a scale | -35.7 (20.3) | -29.2 (21.7)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0087, ANOVA

16. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Monovisc® (PP)
Description: Mean change in knee pain from baseline to 3 weeks as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Monovisc® group (PP population). The WOMAC Pain Score is a validated visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 3 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 137 | 135
score on a scale | -41.3 (19.2) | -35.3 (22.0)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0154, ANOVA

17. Secondary Outcome: OMERACT-OARSI Responder Index Comparing Cingal® to Saline (PP)
Description: The post treatment Responder Rate comparing Cingal® and Saline at 12 weeks is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index (PP population). The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder. The criteria for response are (1) improvement in pain or physical function ≥50% and an absolute change ≥20 mm; or (2) improvement of ≥20% with an absolute change ≥10 mm in at least two of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome.
Time Frame: 12 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Number; unit: percentage of subjects
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 137 | 63
percentage of subjects | 92.8 | 83.6
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0227, ANOVA

18. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Saline (PP)
Description: Mean change from baseline to 12 weeks in the Patient Global Assessment (PGA) comparing the Cingal® and Saline arms (PP population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 12 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 137 | 63
score on a scale | -37.8 (1.5) | -26.0 (2.6)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority or Other; p = 0.0002, ANOVA

19. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Monovisc® (PP)
Description: The post treatment Responder Rate comparing Cingal® and Monovisc® at 1 week is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index (PP population). The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder. A higher percentage of subjects responding indicates a better outcome.
Time Frame: 1 Week
Population: Per Protocol (PP) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 136 | 135
score on a scale | -33.7 (22.3) | -27.1 (22.2)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0148, ANOVA

20. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Monovisc® (PP)
Description: Mean change from baseline to 3 weeks in the Patient Global Assessment (PGA) comparing the Cingal® and Monovisc® arms (PP population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 3 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 137 | 135
score on a scale | -39.2 (20.9) | -32.4 (22.7)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0113, ANOVA

21. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score Comparing Cingal® to Saline. (PP)
Description: Mean change in knee pain from baseline to 26 weeks as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score comparing the Cingal® group to the Saline group (PP population). The WOMAC Pain Score is a validated 100mm visual analog scale from 0 mm = no pain to 100 mm = highest pain level. A negative number for the difference from baseline indicates reduction in pain. A greater negative difference from baseline means a better outcome.
Time Frame: 26 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 134 | 62
score on a scale | -41.2 (1.4) | -32.4 (2.3)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0016, ANOVA

22. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Saline (PP)
Description: Mean change from baseline to 12 weeks in the Evaluator Global Assessment comparing the Cingal® and Saline arms (PP population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 12 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 137 | 63
score on a scale | -37.7 (1.5) | -28.4 (2.9)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0056, ANOVA

23. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® and Monovisc® (PP).
Description: Mean change from baseline to 1 week in the Evaluator Global Assessment comparing the Cingal® and Monovisc® arms (PP population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 1 Week
Population: Per Protocol (PP) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 136 | 135
score on a scale | -32.9 (19.2) | -26.5 (19.2)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0095, ANOVA

24. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Monovisc® (PP)
Description: Mean change from baseline to 3 weeks in the Evaluator Global Assessment comparing the Cingal® and Monovisc® arms (PP population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 3 Week
Population: Per Protocol (PP) Population to compare Cingal® group to Monovisc® group. Saline group is analyzed separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®)
Number analyzed (Participants) | 137 | 135
score on a scale | -38.6 (20.4) | -32.0 (20.9)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Hyaluronic Acid (Monovisc®); Test type: Superiority; p = 0.0136, ANOVA

25. Secondary Outcome: Patient Global Assessment (PGA) Comparing Cingal® to Saline (PP)
Description: Mean change from baseline to 26 weeks in the Patient Global Assessment (PGA) comparing the Cingal® and Saline arms (PP population). The PGA is completed by the subject answering the question "Considering all the ways the osteoarthritis in your STUDY knee affects you, what is your assessment of how much your STUDY knee is bothering you today?" The PGA is scored on a 100mm visual analog scale, where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates an improvement in the patient assessment. A greater negative difference means a better outcome.
Time Frame: 26 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 134 | 62
score on a scale | -38.6 (1.6) | -27.0 (2.7)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0005, ANOVA

26. Secondary Outcome: Evaluator Global Assessment Comparing Cingal® to Saline (PP)
Description: Mean change from baseline to 26 weeks in the Evaluator Global Assessment comparing the Cingal® and Saline arms (PP population). The Evaluator Global Assessment is completed by the Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a visual analog scale where 0 = the patient is not bothered, to 100 mm = the patient is bothered to the highest degree. A negative number for the difference from baseline indicates improvement in the assessment. A greater negative difference means a better outcome.
Time Frame: 26 Weeks
Population: Per Protocol (PP) Population to compare Cingal® group to Saline group. Monovisc® group is analyzed separately.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Saline
Number analyzed (Participants) | 134 | 62
score on a scale | -39.1 (1.5) | -29.8 (2.9)
Statistical Analysis 1: Comparison: Hyaluronic Acid and TH (Cingal®) vs Saline; Test type: Superiority; p = 0.0059, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected at baseline, and at 1, 3, 6, 12, 18 and 26 week follow-up visits.
Description: Definitions used are in accordance with clinicaltrials.gov definitions
Arm/Group | Hyaluronic Acid and TH (Cingal®) | Hyaluronic Acid (Monovisc®) | Saline
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/150 | 0/69
Serious Adverse Events (participants affected / at risk) | 2/149 | 0/150 | 3/69
Other Adverse Events (participants affected / at risk) | 36/149 | 37/150 | 12/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronic Acid and TH (Cingal®) (N=149) | Hyaluronic Acid (Monovisc®) (N=150) | Saline (N=69)
Benign Neoplasm of Adrenal Gland (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Herniated Disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Post-Laminectomy Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mania Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Facial Nerve Damage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronic Acid and TH (Cingal®) (N=149) | Hyaluronic Acid (Monovisc®) (N=150) | Saline (N=69)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 8 (8) | 8 (8) | 2 (2)
Migrane (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
VIIth nerve injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No